CLINICAL TRIAL: NCT03569735
Title: Nanshan Elderly Cohort Study：a Community-based Prospective Cohort Study in Nanshan， Shenzhen Residents
Brief Title: Nanshan Elderly Cohort Study
Acronym: NECS
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shenzhen Nanshan Center for Chronic Disease Control (Unknown)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Other Study IDs: 2017005
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus; Cardiovascular Diseases; Stroke; Obesity; Metabolic Syndrome; Sarcopenia; Chronic Kidney Disease; Cancer; Death
Keywords: Prospective Cohort Study; Nutrition; Chronic diseases; Nanshan; Chinese
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Stroke; Obesity; Metabolic Syndrome; Sarcopenia; Renal Insufficiency, Chronic; Neoplasms; Death; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Overnight fasting blood sample, early morning first-void urine sample and faeces samples will be collected at baseline and follow-up。
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: The Nanshan Elderly Cohort Study (NECS) aims to investigate the nutritional, as well as other environmental and genetic factors of chronic diseases, such as cardio-metabolic diseases.

Study design: NECS is a community-based prospective cohort study. Participants: About 10000-20000 apparently healthy residents, living in Nanshan， Shenzhen (South China) for >5 years, aged ≥ 65 years, will be recruited between 2018 and 2019.

Visits and Data Collection: Participants will be followed up approximately every 3 years by invited to the Community Healthcare Service Centre. At each survey, face-to-face interviews, anthropometric measurements, ultrasonography examination, electrocardiogram test and specimen collection will be conducted.

Key variables:

1. Face-to-face interviews: Structured questionnaires will be used to collect the participants' socio-demographic characteristics, lifestyles, habitual dietary intake, physical activity, history of chronic diseases, use of supplements and medications, family history, psychological health and cognitive function.
2. Physical examinations: Anthropometric measurements, blood pressure tests, handgrip strength, and usual gait speed.
3. Ultrasonography examinations: Ultrasonography examination will be performed to determine carotid artery intima-media thickness and plaque, fatty liver.
4. Electrocardiogram test: Electrocardiogram test is to obtain information about the structure and function of the heart.
5. Specimen collections: Overnight fasting blood sample, early morning first-void urine sample and faeces samples will be collected and stored at -80°C till tests.
6. Laboratory tests:

   1. Blood tests: Metabolic syndrome-related indices; nutritional indices; inflammatory markers; sexual hormones; genetic markers.
   2. Urinary tests: Flavonoids and flavones, minerals, creatinine and renal function related markers.
   3. Fecal test: Gut microbiota and related metabolites.
7. Morbidity and mortality: Relevant data will be also retrieved via local multiple Health information systems.
8. Others: Many other laboratory tests or instrument tests will be developed depended on needs and resources in future.

DETAILED DESCRIPTION:
Objective: The Nanshan Elderly Cohort Study (NECS) aims to investigate the nutritional, as well as other environmental and genetic factors of chronic diseases, such as hypertension, type 2 diabetes mellitus, cardiovascular diseases, stroke, obesity, metabolic syndrome, chronic kidney disease, cancer and sarcopenia.

Study design: NECS is a community-based prospective cohort study. Participants: Healthy residents who had lived in Nanshan， Shenzhen (South China) for >5 years, aged ≥ 65 years are eligible. Participants would be excluded if they are confirmed to have serious chronic diseases, such as cardiovascular disease, liver or renal failure, or cancer. About 10000-20000 apparently healthy residents will be recruited between 2018 and 2019.

Visits and Data Collection: Participants will be followed up approximately every 3 years by invited to the Community Healthcare Service Centre. At each survey, face-to-face interviews, anthropometric measurements, ultrasonography examinations, electrocardiogram test and specimen collection will be conducted.

Key variables:

1. Face-to-face interviews: Structured questionnaires will be used to collect the participants' socio-demographic characteristics (e.g., age, sex and household income, education level), lifestyles (smoking, passive smoking, alcohol and tea drinking), habitual dietary intake (a 62-item quantitative food frequency questionnaire), physical activity, history of chronic diseases, use of supplements and medications, family history, psychological health (Self-Rating Anxiety Scale, SAS), social support and participation, cognitive function (Mini-Mental State Examinations, MMSE);
2. Physical examinations: Anthropometric measurements (weight, height, waist, hip and neck circumference, etc.), blood pressure tests, handgrip strength, and usual gait speed.
3. Ultrasonography examinations: Ultrasonography examination of the carotid artery and upper abdominal organs (e.g., liver and kidney) will be performed to determine carotid artery intima-media thickness and plaque, fatty liver.
4. Electrocardiogram test: Electrocardiogram test is to obtain information about the structure and function of the heart.
5. Specimen collections: Overnight fasting blood sample will be collected and separated into serum, plasma, red blood cell and leukocyte within two hours. Early morning first-void urine sample and faeces samples will be collected. All specimens will separated and stored at -80°C till tests.
6. Laboratory tests:

   1. Metabolic syndrome-related indices: Fasting serum lipid profile (e.g., cholesterol, triglycerides, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol), diabetes-related indices (e.g., glucose, glycated hemoglobin, fructosamine and insulin), uric acid and creatinine;
   2. Nutritional indices: Serum concentrations of carotenoids, erythrocyte fatty acids, serum minerals, folate, betaine, choline, TMAO, and vitamin D, etc.
   3. Inflammatory markers (e.g., hsCRP, RBP4，IL-6, TNF-a)
   4. Sexual hormones (e.g., testosterone, SHBG)
   5. Genetic markers
   6. Urinary tests: Flavonoids and flavones, minerals, creatinine and renal function related markers.
   7. Fecal test: Gut microbiota and related metabolites.
7. Morbidity and mortality: Relevant data will be also retrieved via local multiple Health information systems.
8. Others: Many other laboratory tests or instrument tests will be developed depended on needs and resources in future.

Statistical analysis: Cox proportional hazards models or logistic regression models will be used to estimate the risk of exposures on categorical outcomes. Path analysis also will be used to assess the potential mediating effects in the causal pathway between exposures and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 65 years;
* Living in Nanshan, Shenzhen for at least 5 years;
* Chinese.

Exclusion Criteria:

* Had a history of hospital-confirmed diabetes, failure(s) of heart, liver, or kidney, cancer, CVD events;
* On special diet due to a disease or weight control;
* Mental and physical disability;
* Likely to move to other city within 5 years;
* Did not want to attend any one item of the survey or sample collection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The participants who meet the inclusion and exclusion criteria will be recruited from all communities of Nanshan, Shenzhen by face-to-face communication.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-05-26 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes mellitus | Up to 10 years
  The investigators will also track for occurrence of diabetes mellitus by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Shenzhen Center for Disease Control and Prevention and Health Insurance Bureau. All cases will be verified by medical record reviews.
Cardiovascular diseases (occurrence of cardiovascular diseases) | Up to 10 years
  The investigators will track for occurrence of cardiovascular diseases by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Shenzhen Center for Disease Control and Prevention, and Health Insurance Bureau. All cases will be verified by medical record reviews.
Stroke (occurrence of stroke) | Up to 10 years
  The investigators will track for occurrence of stroke by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Shenzhen Center for Disease Control and Prevention, and Health Insurance Bureau. All cases will be verified by medical record reviews.
Cognitive disorder (occurrence of cognitive disorder) | Up to 10 years
  The investigators will track for occurrence of cognitive disorder by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Shenzhen Center for Disease Control and Prevention, and Health Insurance Bureau. All cases will be verified by medical record reviews.

SECONDARY OUTCOMES:
Metabolic syndrome | Up to 10 years
  The investigators will measure metabolic syndrome-related indices at each visit (per every 3 years), the investigators can analysis the incidence of metabolic syndrome.
Change lipid profile | Up to 10 years
  The investigators will measure fasting lipid profile (e.g., cholesterol, triglycerides, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol) at each visit, and analyse the change of these indices.
Handgrip strength | Up to 10 years
  The investigators will measure the handgrip strength, which will be used to diagnose sarcopenia according to definition recommended by Asian Working Group for Sarcopenia (AWGS): cutoff values for handgrip strength (<26 kg for men and <18 kg for women).
Usual gait speed | Up to 10 years
  The investigators will measure the usual gait speed., which will also be used to diagnose sarcopenia according to definition recommended by Asian Working Group for Sarcopenia (AWGS): cutoff values for usual gait speed (<0.8 m/s).

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Chen, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Department of Non-communicable Disease Prevention and Control, Shenzhen Nanshan Center for Chronic Disease Control, Shenzhen, Guangdong
  - Department of Medical Statistics & Epidemiology, School of Public Health, Sun Yat-sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No